CLINICAL TRIAL: NCT03356639
Title: A Phase 1 Randomized, 2-way, Crossover Study to Assess the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of ASP6981 in Patients With Schizophrenia
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of ASP6981 in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6981-CL-0004
Record Dates: First submitted 2017-11-28; First posted 2017-11-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; ASP6981; Safety; Phase 1
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ASP6981 50 mg, then matching Placebo (Experimental): Participants in Sequence AB will first receive ASP6981 capsules orally (50 mg) during period 1. After a 14-day washout period, participants receive matching placebo during period 2. Participants will receive ASP6981 capsules or matching placebo capsules every 12 hours on days 1 through 14 (only in the morning of day 14) of period 1 and 2. On days 1 and 14 of period 1 and 2, ASP6981 or matching placebo will be administered under fasting conditions.
  Interventions: Drug: ASP6981; Drug: Placebo
- Matching Placebo, then ASP6981 50 mg (Experimental): Participants in Sequence BA will first receive matching placebo capsules orally during period 1. After a 14-day washout period, participants receive ASP6981 capsules (50 mg) during period 2. Participants will receive matching placebo or ASP6981 capsules every 12 hours on days 1 through 14 (only in the morning of day 14) of period 1 and 2. On days 1 and 14 of period 1 and 2, matching placebo or ASP6981 will be administered under fasting conditions.
  Interventions: Drug: ASP6981; Drug: Placebo
- ASP6981 135 mg, then matching Placebo (Experimental): Participants in Sequence CD will first receive ASP6981 capsules orally (135 mg) during period 1. After a 14-day washout period, participants receive matching placebo during period 2. Participants will receive ASP6981 capsules or matching placebo every 12 hours on days 1 through 14 (only in the morning of day 14) of period 1 and 2. On days 1 and 14 of period 1 and 2, ASP6981 or matching placebo will be administered under fasting conditions.
  Interventions: Drug: ASP6981; Drug: Placebo
- Matching Placebo, then ASP6981 135 mg (Experimental): Participants in Sequence DC will first receive matching placebo capsules orally during period 1. After a-14 day washout period, participants receive ASP6981 (135 mg) during period 2. Participants will receive matching placebo or ASP6981 capsules every 12 hours on days 1 through 14 (only in the morning of day 14) of period 1 and 2. On days 1 and 14 of period 1 and 2, matching placebo or ASP6981 will be administered under fasting conditions.
  Interventions: Drug: ASP6981; Drug: Placebo

INTERVENTIONS:
Drug: ASP6981 — Oral
Drug: Placebo — Oral

SUMMARY:
The primary purpose is to evaluate the safety and tolerability of ASP6981 in participants with schizophrenia.

Also primary purpose is to evaluate the pharmacodynamics of ASP6981 in participants with schizophrenia as measured by cognitive function and neurophysiological biomarkers.

The secondary purpose of this study is to evaluate the pharmacokinetics of ASP6981 in participants with schizophrenia.

DETAILED DESCRIPTION:
This study will evaluate ASP6981 in stable participants with schizophrenia on stable doses of up to 2 second generation antipsychotic drugs for at least 2 months prior to screening. Participants will be enrolled and randomized into 1 of 4 treatment sequences: AB, BA, CD, DC.

Screening period: After a screening period of up to 29 days prior to study drug administration, eligible participants will be admitted to the clinical unit on day -3.

Investigational period: Enrolled participants will be randomized to receive either ASP6981 or Placebo first and then will be crossed over to receive the opposite intervention. The study will consist of two treatment periods of 14 days separated by a washout period of 14 days. Participants will be discharged from the clinical unit on day 15 for the washout period. Washout may be extended up to a maximum of 21 days depending on the participant's availability.

Follow up: Participants will return to the clinical unit for an End of Study Visit (ESV) on day 28 of period 2 or, if the participant terminated early from the study, 14 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria.
* Subject is considered operationally stable if the subject has a low to moderate positive symptom score and moderate negative symptom score on the PANSS (Positive and Negative Syndrome Scale): no more than moderate rating on more than 2 PANSS items P1, P2, P3, P5, P6; no more than moderate severity rating for the negative items, N1, N2, N3, N4, N5, N6, N7; total PANSS score no more than 80.
* Subject must be in ongoing maintenance antipsychotic therapy (i.e., second generation antipsychotics other than clozapine oral or depot), on a stable (less than or equal to 25% change in dose) medication treatment regimen (approved oral or depot formulations of risperidone, quetiapine, olanzapine, ziprasidone, brexpiprazole, aripiprazole, paliperidone or lurasidone; up to 2 permitted on condition that the second medication is not required to control treatment resistance or intractable psychotic symptoms) for more than or equal to 2 months for oral formulations or more than or equal to 3 months for depot formulations prior to screening, including concomitant psychotropic medications, such as, trazodone and zolpidem for sleep.
* Subject has a body mass index (BMI) range of 18.5 to 40.0 kg/m2, inclusive, and weighs at least 50 kg.
* Subject has a negative urine drug screen for drugs of abuse.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* A sexually active male subject with female partner(s) who are of childbearing potential is eligible if:

  * The male subject agrees to use a male condom starting at screening and continue throughout the study period and for 90 days after the final study drug administration.
  * The male subject has not had a vasectomy or is not sterile, as defined above, their female partner(s) is utilizing 1 form of highly effective birth control starting at screening and continuing throughout study treatment and for 90 days after the male subject receives their final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until completion of the ESV.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP6981 or any components of the formulation used.
* Subject has had previous exposure with ASP6981.
* Subject has a history of heavy smoking (use more than 40 cigarettes/2 packs per day) or a user of nicotine replacement therapy (includes nicotine patches, Chantix or similar therapeutic agents) in the past 3 months prior to admission to the clinical unit (day -3).
* Subject has a history of suicide attempt or suicidal behavior within 2 years prior to screening. Any suicidal ideation that meets criteria at a level of 4 or 5 by using C-SSRS within the last 3 months or who is at significant risk to commit suicide will be excluded.
* Subject has any clinically significant liver chemistry test result (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma glutamyl transferase, total bilirubin [TBL]) or a result greater than 1.5 x greater than upper limit of normal (ULN). In such a case, the assessment may be repeated once.
* Subject has any history of allergic conditions deemed clinically significant.
* Subject has any history or evidence of any clinically significant cardiovascular, gastro-intestinal endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric (other than schizophrenia or schizoaffective disorder), renal and/or other major disease or malignancy.
* Subject has a history of being diagnosed with moderate or severe tardive dyskinesia, bipolar disorder, major depressive disorder, personality disorders, neuroleptic malignancy syndrome or anxiety disorder.
* Subject has any clinically significant abnormality of the physical examination, ECG and protocol-defined clinical laboratory tests.
* Subject has a mean pulse lower than 40 or greater than 100 bpm; resting systolic blood pressure (SBP) lower than 90 or greater than 180 mmHg, or a resting diastolic blood pressure (DBP) greater than 100 mmHg at screening and on day -3 (measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically). If the mean blood pressure exceeds the limits above, 1 additional triplicate can be taken at screening and on day -3.
* Subject has a mean QT interval using Fridericia's correction (QTcF) of greater than 450 ms (for male subjects) and greater than 470 ms (for female subjects). If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken at screening and on day -3.
* Subject uses any prescribed (including current treatment with anticholinergic medications such as benztropine, biperiden, procyclidine, and trihexyphenidyl) or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., valerian) in the 2 weeks prior to study drug administration until the ESV, except for:

  * Approved second generation antipsychotics (risperidone, quetiapine, olanzapine, ziprasidone, brexpiprazole, aripiprazole, paliperidone or lurasidone), or
  * Approved intermittent use of short-acting hypnotic agents trazodone or zolpidem (no less than 12 hours prior to dosing), or
  * Approved intermittent use of anticholinergic compounds, or
  * Approved use of concomitant medication for the treatment of hypertension, hyperlipidemia or diabetes mellitus, or
  * Occasional use of acetaminophen (up to 2 g/day), or
  * Hormonal contraceptives, or
  * Hormone replacement therapy.
* Subject has a history of consuming more than: 14 units of alcoholic beverages per week for male subjects or 7 units of alcoholic beverages per week for female subjects within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol or drugs of abuse at screening or at admission to the clinical unit (day -3 of period 1). Subject tests positive for benzodiazepines at admission to the clinical unit (day -3 of period 1).
* Subject who is unable to refrain from smoking or drinking coffee for 3 hours prior to the Cogstate and EEG testing.
* Subject has used any strong CYP3A inhibitors (e.g., but not limited to: boceprevir, clarithromycin, conivaptan, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, voriconazole) and/or has consumed grapefruit, grapefruit-containing products, Seville orange or Seville orange-containing products within 72 hours prior to admission to the clinical unit (day -3 of period 1).
* Subject regularly uses any inducer of CYP3A metabolism (e.g., but not limited to: carbamazepine, phenytoin, rifampin, St. John's Wort, bosentan, efavirenz, etravirine, modafinil, nafcillin, amprenavir, aprepitant, armodafinil, clobazamechinacea, pioglitazone, prednisone, rufinamide, vemurafenib) in the 3 months prior to admission to the clinical unit (day -3 of period 1).
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies or human immunodeficiency virus antibodies type 1 or 2.
* Subject who has had electroconvulsive therapy within the 6 months prior to screening.
* Subject has a history of seizures or of a condition with risk of seizures; as an exception, a history of 1 febrile seizure in childhood will not exclude a subject.
* Subject has a history of head injury with clinically significant sequelae.
* Subject experienced an acute exacerbation of schizophrenia requiring hospitalization or an increase in antipsychotic medication (with reference to drug or dose) within the last 2 months prior to screening.
* Subject has hearing loss, is unable to detect 1000 Hz tones presented at 40 dB.
* Subject has a condition which makes the subject unable to complete or perform the EEG assessments defined in the study (e.g., dreadlocks), during the study screening period.
* Subject has a history of spine surgery (with intact dura mater) in the past year and/or a history of brain and/or spinal cord injury.
* Subject has a condition which makes the subject unable to complete the study cognitive assessments defined in the study, during the study screening period.
* Subject has any condition, which makes the subject unsuitable for study participation.
* Subject has participated in any study or has been treated with any investigational drugs within 28 days or 5 half-lives whichever is longer, prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by nature, frequency and severity of adverse events (AEs) | Up to End of Study (up to a maximum of 65 days)
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Number of participants with vital signs abnormalities and/or adverse events related to treatment | Up to End of Study (up to a maximum of 65 days)
  Number of participants with potentially clinically significant vital sign values.
Number of participants with laboratory value abnormalities and/or adverse events related to treatment | Up to End of Study (up to a maximum of 65 days)
  Number of participants with potentially clinically significant laboratory values.
Safety and tolerability assessed by 12-lead electrocardiogram (ECG) | Up to End of Study (up to a maximum of 65 days)
  Routine 12 lead ECGs will be performed after the participant has been in a supine position for at least 5 minutes.
  Any clinically significant adverse changes on the ECG will be reported as (serious) Adverse Event.
Safety and tolerability assessed by C-SSRS | Up to 50 days
  C-SSRS: Columbia - Suicide Severity Rating Scale. The C SSRS is a rating scale that assesses the full spectrum of suicidality: suicide ideation, intensity of ideation, suicidal behaviors and actual attempts.
Safety and tolerability assessed through metabolic parameter: waist circumference | Up to End of Study (up to a maximum of 65 days)
  Waist circumference will be summarized by ASP6981 treatment group and pooled placebo.
Safety and tolerability assessed through metabolic parameter: lipid panel | Up to End of Study (up to a maximum of 65 days)
  Lipid panel will be summarized by ASP6981 treatment group and pooled placebo.
Safety and tolerability assessed through metabolic parameter: glucose level | Up to End of Study (up to a maximum of 65 days)
  Glucose level will be summarized by ASP6981 treatment group and pooled placebo.
Safety and tolerability assessed by weight | Up to End of Study (up to a maximum of 65 days)
  Weight to be summarized by ASP6981 treatment group and pooled placebo.
Safety and tolerability assessed for movement disorder using AIMS | Up to 50 days
  AIMS: Abnormal Involuntary Movement Scale. The AIMS aids in the early detection of tardive dyskinesia as well as providing a method for on going surveillance. The AIMS is a checklist and uses a 5 point rating scale for recording scores for 7 body areas: face, lips, jaw, tongue, upper extremities, lower extremities and trunk.
Safety and tolerability assessed for movement disorder using BARS | Up to 50 days
  BARS: Barnes Akathisia Rating Scale. The BARS is a rating scale that is used to assess the severity of drug induced akathisia.
Safety and tolerability assessed for movement disorder using SAS | Up to 50 days
  SAS: Simpson Angus Scale. The SAS is a 10 item scale used to rate adverse neurological effects of antipsychotic medications more broadly. It involves direct observation and a brief neurological examination. Rating requires the investigator to observe the participant's gait and check for tremor, excessive salivation and rigidity in the arms, shoulder and neck. Each item is rated from 0 to 4 and a total score can be obtained.
Pharmacodynamics (PD) of ASP6981 assessed through Cogstate: general composite score of executive function and memory cognitive testing | Day 14: period 1 and 2
  Cogstate testing composed by Groton Maze Learning, One Back, One Card and International Shopping List tests: specific Cogstate's panels for schizophrenia.
PD of ASP6981 assessed through electroencephalogram (EEG): electrophysiological measures of P300 (P3a, P3b) and Mismatch Negativity (MMN) | Day 14: period 1 and 2
  EEG will be recorded after cognitive testing.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP6981 and its metabolites, if necessary (plasma): Tmax | Day 1 and day 14: period 1 and 2
  Tmax: time of maximum concentration
PK of ASP6981 and its metabolites, if necessary (plasma): Cmax | Day 1 and day 14: period 1 and 2
  Cmax: maximum concentration
PK of ASP6981 and its metabolites, if necessary (plasma): AUC12 | Day 1: period 1 and 2
  AUC12: Area under the concentration time curve from the time of dosing to 12 hours postdose
PK of ASP6981 and its metabolites, if necessary (plasma): Ctrough | Day 7 and day 14: period 1 and 2 and day 13 of period 2
  Ctrough: Concentration immediately prior to dosing at multiple dosing
PK of ASP6981 and its metabolites, if necessary (plasma): AUCtau | Day 14: period 1 and 2
  AUCtau: Area under the concentration time curve from the time of dosing to the start of the next dosing interval
PD of ASP6981 assessed through Cogstate: composite score of attention cognitive testing | Day 14: period 1 and 2
  Cogstate testing composed by Detection Test and Identification.
PD of ASP6981 assessed through EEG: electrophysiological measures of Auditory Steady State Response (ASSR), N100, P200 and resting state | Day 14: period 1 and 2
  EEG will be recorded after cognitive testing.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (2):
- United States (2):
  - Cctmg/Parexel, Glendale, California
  - Community Clinical Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=331